CLINICAL TRIAL: NCT06382285
Title: The Effect of a Prolonged Peripheral Nerve Block (Utilazing Continuous Adductor Canal Block on the Level of Pain After a Knee Replacement Surgery
Brief Title: The Effect of a Prolonged Peripheral Nerve Block on the Level of Pain After a Knee Replacement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Zoya Haitov Ben Zikri, Director of the anesthesia department, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0206-22-ASF
Record Dates: First submitted 2023-09-07; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Knee Replacement Surgery

STUDY DESIGN:
Intervention Model Description: The study will include 50 patients who underwent a knee replacement surgery, who will be randomized to 2 groups. 6 hours after surgery the two groups will be connected to a prolonged block pump. One group will receive the peripheral block ropivacaine 0.2% according to the protocol of 8-10 cc per hour up to 24 hours after surgery. The second group will receive saline according to the same protocol
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): ropivacaine (Naropin) 0.2% according to a protocol 8-10 cc per hour up to 24 hours after the surgery
  Interventions: Drug: Continues peripheral block
- Control group (Placebo Comparator): Saline according to a protocol 8-10 cc per hour up to 24 hours after the surgery
  Interventions: Drug: Continues peripheral block

INTERVENTIONS:
Drug: Continues peripheral block — ropivacaine (Naropin) 0.2% according to a protocol 8-10 cc per hour up to 24 hours after surgery
  Other Names: Treatment group

SUMMARY:
The aim of this study is to examine the effect of a prolonged peripheral nerve block (utilizing continuous adductor canal block) on the level of pain after a knee replacement surgery

DETAILED DESCRIPTION:
Knee replacement surgery is one of the common orthopedic surgeries for the treatment of chronic knee pain. The period after knee replacement surgery is accompanied by moderate to severe pain that affects the patient's ability to quickly return to function. Peripheral nerve blockers and analgesia of different types, administered as part of the anesthesia process, are optimal in controlling pain after surgery. After the surgery, the patients are admitted in the orthopedic inpatient department for 2-3 days on average after surgery for follow-up and early physical therapy necessary to achieve good results and return the patient to full function as soon as possible. The level of pain greatly affects the success rate of the patient's rehabilitation. Thus, since the duration of peripheral nerve block activity does not exceed 8-16 hours on average, it is suggested to treat the patients with a prolonged peripheral nerve block (utilizing continuous adductor canal block) for 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients between the ages of 18 and 80 who have signed an informed consent form.
* ASA is less than 3
* Spinal anesthesia

Exclusion Criteria:

* Patients with sensitivity to the anesthetic.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain level | during hospitalization (1-2 days)
  Documentation of pain level during the hospitalization days every 12 hours (on a scale of 1-10)
Analgesic use | during hospitalization (1-2 days)
  Documentation of pain level during the hospitalization days every 12 hours (on a scale of 1-10).
  Documentation of analgesic administration in hospitalization.

SECONDARY OUTCOMES:
Physiotherapy | during hospitalization (1-2 days)
  Documentation of the execution of a full or partial physical therapy program

IPD SHARING:
Plan to Share IPD: No